CLINICAL TRIAL: NCT02887313
Title: Totally Neoadjuvant Chemoradiation Therapy With mFOLFOX6 in Locally Advanced Rectal Cancer: A Real World Study
Brief Title: FOLFOX6 Totally Neoadjuvant Chemoradiation Therapy in Locally Advanced Rectal Cancer: A Real World Study
Acronym: FOTAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU11
Record Dates: First submitted 2016-08-27; First posted 2016-09-02 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Neoadjuvant chemoradiation therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Locally advanced rectal cancer (Experimental): Locally advanced rectal cancer receiveing total neoadjuvant treatment
  Interventions: Drug: mFOLFOX6; Radiation: Radiotherapy

INTERVENTIONS:
Drug: mFOLFOX6 — Patients receive mFOLFOX6 for 4 cycles during neoadjuvant radiotherapy, and after CRT, another 4 cycles of mFOLFOX6 would be given before surgery.
  Other Names: fluorouracil; oxaliplatin; Leucovorin
Radiation: Radiotherapy — Patietns received preoperative radiotherapy, 1.8-2.0GY/23-25F

SUMMARY:
Preoperative 5FU based chemoradiotherapy is still the standard of treatment for locally advanced rectal cancer. About 15-20% of patients would achieve pathologic complete response (pCR) after neoadjuvant CRT, and the survival outcome was much better than that of non-pCR. Total neoadjuvant treatment had been evaluated a lot in recent years, including induction chemotherapy or consolidation chemotherapy, or concurrent chemoradiotherapy. We aimed to evaluated the safety and efficacy of total neoadjuvant treatemnt in locally advanced rectal cancer.

DETAILED DESCRIPTION:
Preoperative 5FU based chemoradiotherapy is still the standard of treatment for locally advanced rectal cancer. About 15-20% of patients would achieve pathologic complete response (pCR) after neoadjuvant CRT, and the survival outcome was much better than that of non-pCR. However, distant metastasis would occur in about 30% of patients even after CRT. To improve the survival of rectal cancer patients, we hope to improve the pCR rate. In our previous FOWARC study, mFOLFOX6 with radiation had the pCR rate of 27.5%. It had been reported that adding FOLFOX after neoadjuvant chemo radiation in locally advanced rectal cancer would improve pCR rate. Nowadays, induction or consolidation chemotherapy or concurrent chemoradiotherapy had been used in clincal practice. Here, we are going to evaluate the safety and efficacy of total neoadjuvant therapy in real world.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the rectum
* Age: 18-70 years old
* Signed informed consent; able to comply with study and/or follow- up procedures
* Stage of the primary tumor may be determined by ultrasound or MRI
* Stage II (T3-4, N0 [N0 is defined as all imaged lymph nodes < 1.0 cm]) OR stage III (T1-4, N1-2 [with the definition of a clinically positive lymph node being any node ≥ 1.0 cm]
* Tumor palpable by digital rectal exam OR accessible by proctoscope or sigmoidoscope
* Distal border of the tumor must be located < 12 cm from the anal verge
* Tumor amenable to curative resection
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:
* Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥ 9g/ dL.
* Total bilirubin ≤1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
* Alkaline phosphatase limit ≤ 5x ULN.
* Amylase and lipase ≤ 1.5 x the ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.
* No renal disease that would preclude study treatment or follow-up
* ECOG status: 0～1

Exclusion Criteria:

* Hypersensitivity to fluorouracil, oxaliplatin or irinotecan.
* No More than 4 weeks since prior participation in any investigational drug study
* More than 4 weeks since prior participation in any investigational drug study
* Clear indication of involvement of the pelvic side walls by imaging
* With distant metastasis
* History of invasive rectal malignancy, regardless of disease-free interval
* Fertile patients must use effective contraception
* Uncontrolled hypertension
* Cardiovascular disease that would preclude study treatment or follow-up
* Lack of upper gastrointestinal tract integrity or malabsorption syndrome，active upper gastrointestinal tract bleeding
* Synchronous colon cancer
* Pregnant or nursing, Fertile patients do not use effective contraception
* Other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
* No psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation
* patients refused to signed informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-05 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 2 years
  The pathologic outcome after neoadjuvant CRT showed no tumor residual.

SECONDARY OUTCOMES:
Safety and compliance of treatment | 2 years
  The adverse events after total neoadjuvant treatment
The ratio of tumor downstaging to stage 0 and stage I | 2 years
  Tumor downstaging from stage II or III to pathologic complete response (stage 0) and stage I
Disease free survival | 3 years
  3 years recurrence free survival of this group of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Gastrointestinal Hospital, Sun Yatsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes